CLINICAL TRIAL: NCT06436755
Title: Effect of Serratus Anterior Plane Block and Transthoracic Plane Block Combination on Postoperative Analgesia From Pectus Surgery
Brief Title: Serratus Anterior Plane Block and Transthoracic Plane Block in Pectus Surgery
Status: Recruiting | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Cansu KILINC BERKTAS, Specialist MD, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2024-271
Record Dates: First submitted 2024-05-15; First posted 2024-05-31 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-05

CONDITIONS: Pectus Excavatum
Keywords: Transversus thoracic muscle plane block; postoperative analgesia; pectus excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serratus anterior plane block (SAP) group: Patients who underwent serratus anterior plane block
  Interventions: Procedure: no intervention,this is a observational studies
- Serratus anterior plane block (SAP) and Transversus thoracic plane block (TTP) group: Patients who underwent Serratus anterior plane block (SAP) and Transversus thoracic plane block (TTP) group
  Interventions: Procedure: no intervention,this is a observational studies

INTERVENTIONS:
Procedure: no intervention,this is a observational studies — no intervention,this is a observational studies

SUMMARY:
The most important problem in the postoperative period in patients scheduled for pectus deformity correction surgery is pain. Due to the catastrophic neurological complications of thoracic epidural analgesia, the tendency towards plane blocks has been increasing in recent years. Serratus Plane Block (SAP Block), performed under ultrasound guidance, is used to treat pain in thoracic surgery. However, whether it has an effect on sternum pain is still controversial and there are not enough studies. Transversus thoracic plane block (TTP Block) provides effective analgesia in sternotomies. For this reason, we aimed to show that the TTP block added to the SAP block will provide more effective analgesia in order to provide adequate analgesia for the pressure and pain sensation of the bars placed on the sternum in pectus surgery.

DETAILED DESCRIPTION:
The most important problem in the postoperative period in patients scheduled for pectus deformity correction surgery is pain. It is very important for patients to start active breathing exercises and mobilize early. Complications develop less frequently in patients who actively breathe and mobilize early. The tolerability of the surgery by the patient and the absence of pain in the postoperative period ensure early discharge . Due to the catastrophic neurological complications of thoracic epidural analgesia, the tendency towards plane blocks has been increasing in recent years. Serratus Plane Block (SAP Block), performed under ultrasound guidance, is used to treat pain in thoracic surgery. However, whether it has an effect on sternum pain is still controversial and there are not enough studies. Transversus thoracic plane block (TTP Block) provides effective analgesia in sternotomies. For this reason, we aimed to show that the TTP block added to the SAP block will provide more effective analgesia in order to provide adequate analgesia for the pressure and pain sensation of the bars placed on the sternum in pectus surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients who will undergo surgery due to pectus deformity All patients over the age of 15 who will be operated on due to pectus deformity

Exclusion Criteria:

* Known allergy to local anesthetics,
* Uncooperative patient,
* The patient who refuses to participate in the study,
* Patients under 18 years of age.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over the age of 15 who will be operated on due to pectus deformity
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2025-11-21 (Estimated)

PRIMARY OUTCOMES:
Effect of Serratus Anterior Plane Block and Transthoracic Plane Block Combination on Postoperative Analgesia in Pectus Surgery | postoperative 48 hours
  Serratus Plane Block (SAP Block), performed under ultrasound guidance, is used to treat pain in thoracic surgery. However, whether it has an effect on sternum pain is still controversial and there are not enough studies. Transversus thoracic plane block (TTP Block) provides effective analgesia in sternotomies. For this reason, TTP block will be added to the SAP block in order to provide adequate analgesia for the pressure and pain sensation of the bars placed on the sternum in pectus surgery.
  The patient's pain score will be evaluated with the Numerical Rating Scale (NRS). Hourly pain scores in the postoperative period are 0./1./4./6./12./18./24./48.
  Additional complications
Postoperative Analgesia in Pectus Surgery | postoperative 48 hours
  Total amount of analgesia for 48 hours,
Postoperative pain in Pectus Surgery | postoperative 48 hours
  Presence of need for additional analgesics,

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam Ve Sakura Şehir Hastanesi, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No